CLINICAL TRIAL: NCT04497831
Title: Determining the Effectiveness of Nebulized Morphine in Treating Dyspnea in Advanced Idiopathic Pulmonary Fibrosis
Brief Title: Morphine for Dyspnea in Pulmonary Fibrosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NKBBN/433/2018; 2019-000662-37 (EudraCT Number)
Record Dates: First submitted 2020-07-25; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, placebo-controlled analysis conducted with crossover arms. The study consists of two treatment periods lasting a total of 5 days: 2 days of nebulization with 0.9% NaCl and 2 days of nebulization with 2.0% morphine hydrochloride solution separated by 1 day intended for elimination of the drug from the body (wash-out). The order of treatment periods (morphine -> placebo, placebo -> morphine) will be randomized for each patient by a hospital pharmacist using online software: Research Randomizer 4.0. The draw will assign the participant to one of two sequences:
  A. 2 days - 0.9% NaCl; 1 day - wash-out; 2 days - morphine hydrochloride. B. 2 days - morphine hydrochloride; 1 day - wash-out; 2 days - 0.9% NaCl
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Drug (Experimental): Morphine hydrochloride
  Interventions: Drug: Morphine hydrochloride
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine hydrochloride — 5 mg milligram(s) per day per two days of dosage
  Arms: Study Drug
Drug: Placebo — Inhalation use
  Arms: Placebo

SUMMARY:
"Determination of the effectiveness of nebulized morphine in the treatment of dyspnea in patients with advanced idiopathic pulmonary fibrosis"

ELIGIBILITY:
Inclusion Criteria:

* IPF diagnosis in accordance with guidelines

  * Period of stable disease
  * Dyspnea rated 3 to 4 in mMRC scale
  * Current non-smoker
  * Other potential causes of breathlessness such as kidney or heart failure optimally treated in the opinion of the principal investigator
  * Able to complete questionnaires and trial assessments
  * Ability to give informed consent
  * If female, must be:

    1. postmenopausal (no menses for 12 months without an alternative medical cause)
    2. sterile
    3. using acceptable contraception and agree to exclude pregnancy with pregnancy test in the beginning of the hospitalization

Exclusion Criteria:

* - other coexisting severe chronic lung diseases
* absolute contraindications to six-minute-walking-test according to

Polish Respiratory Society guidelines:

* < 7-10 days since coronary interventions due to STEMI
* < 24 h since planned coronary intervention
* myocarditis/pericarditis
* symptomatic rhythm and conduction abnormalities
* acute deep vein thrombosis, pulmonary embolism, pulmonary infarction
* decompensated heart failure
* acute infection and other diseases which can significantly impact the test result (eg. severe anemia, acute kidney or liver failure, hypo- or hyperthyroidism, etc)

  - contraindications to morphine hydrochloride:
* previous history of respiratory depression after opioid administration
* previous history of allergic reactions to opioids
* severe ventilation impairment due to e.g. asthmatic state, airway foreign body
* severe kidney or liver failure
* increased intracranial pressure
* head injury
* cerebral edema
* coma
* seizure disorders
* acute alcohol poisoning
* acute abdomen
* acute diarrhea caused by infection or food poisoning;
* patients at risk of paralytic ileus;
* biliary colic;
* phaeochromocytoma;
* simultaneous MAO inhibitor treatment and immediate 2-week period following its discontinuation - ongoing opioid treatment for any indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-21 (Estimated); Primary Completion 2022-09-21 (Estimated); Study Completion 2022-09-21 (Estimated)

PRIMARY OUTCOMES:
The primary end point is a reduction of breathlessness intensity by ≥20 mm at 100 mm visual analogue scale (VAS) after nebulization, during daily, normal activities | Breathlessness during daily, normal activities will be measured with VAS 1 hour before nebulization and 4 hours after
  The primary end point is a reduction of breathlessness intensity by ≥20 mm at 100 mm visual analogue scale (VAS) after nebulization, during daily, normal activities

SECONDARY OUTCOMES:
Secondary end point | Cough and chest pain severity during normal activities will be assessed with VAS 1h before nebulization and 4 hours after Six minute walking test, along with breathlessness, cough and chest pain assessment in VAS, will be performed 1h before nebuli
  Secondary end points are:
  1. reduction of breathlessness intensity by ≥20 mm at 100 mm visual analogue scale (VAS) following six minute walking test (6MWT) performed after nebulization
  2. improvement of 6MWT distance by ≥30 m
  3. reduction of cough severity by ≥17 mm at 100 mm visual analogue scale (VAS) after nebulization, during normal activities
  4. reduction of chest pain severity by ≥19 mm at 100 mm visual analogue scale (VAS) after nebulization, during normal activities
  5. reduction of cough severity by ≥17 mm at 100 mm visual analogue scale (VAS) during six minute walking test (6MWT) performed after nebulization
  6. reduction of chest pain severity by ≥19 mm at 100 mm visual analogue scale (VAS) following six minute walking test (6MWT) performed after nebulization